CLINICAL TRIAL: NCT02965872
Title: Investigating the Learning Effect of Computerized Balance Evaluation System
Brief Title: Learning Effect of Computerized Balance Evaluation System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, PhD, PT, Hacettepe University
Other Study IDs: G0 16/457
Record Dates: First submitted 2016-10-26; First posted 2016-11-17 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Postural Balance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy individuals
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Thirty healthy individuals will be participants of the study. Participants will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass, will be recorded. Postural sway and limits of stability parameters will evaluate with computerized balance evaluation system (BERTEC) for seven times .

DETAILED DESCRIPTION:
Thirty healthy individuals will be participants of the study. Participants will evaluate with the following assessment tools: Demographic datas; age, gender, height, body mass, will be recorded. Postural sway and limits of stability parameters will evaluate with computerized balance evaluation system (BERTEC) for seven times. Every seven evaluations will be repeated while participants in combination of the condition including eyes open, eyes closed, normal surface and perturbated surface.

ELIGIBILITY:
Inclusion Criteria:

* Want to participate

Exclusion Criteria:

* Have passive joint limitation at extremities
* Surgery at last 5 year
* Systemic problems such as neurologic disorders, rheumatoid disorders…
* Another orthopedic anomalies

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy individuals
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Balance evaluation | Initially evaluation at first minute,5 minutes(mns) after the initially evaluation, 10 mns after initially evaluation,15 mns after initially evaluation,20 mns after initially evaluation,25 mns after initially evaluation,30 mns after initially evaluation
  Assessment of ability of protect the balance in conditions including eyes open, eyes closed, normal surface and perturbated surface.

IPD SHARING:
Plan to Share IPD: Undecided